CLINICAL TRIAL: NCT03166514
Title: Pharmacokinetic and Glycemic Response of a Commercially Available Food Bar
Brief Title: Glycemic Response of a Commercial Food Bar
Acronym: NB16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Nutrabolt (Industry)
Responsible Party: Principal Investigator, Richard B. Kreider, Professor, Health & Kinesiology, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB2016-0830D
Record Dates: First submitted 2017-05-05; First posted 2017-05-25 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Glucose and Insulin Response

STUDY DESIGN:
Intervention Model Description: A randomized, cross-over administration of supplements with approximately 5-10 days between testing sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Commercially Available Food Bar (Experimental): 62 g. Fitjoy Bar
  Interventions: Dietary Supplement: Commercially Available Food Bar
- Placebo (Placebo Comparator): 25 g. Dextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Commercially Available Food Bar
  Other Names: Fitjoy Bar
  Arms: Commercially Available Food Bar
Dietary Supplement: Placebo
  Other Names: Dextrose Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the glucose and insulin response to a food bar.

DETAILED DESCRIPTION:
Fitjoy is a commercially available food bar marketed as having a low glycemic index and being relatively high in dietary fiber. The fiber contained within this product is isomalto-oligoshaccaride (IMO) which is a food ingredient with a relative sweetness level equal to approximately 60% of sucrose. Chemically, IMO is a mixture of glucose oligomers with alpha - (1-6) - linkages. To date, no research has been performed on the glycemic response to ingesting IMO in combination with other constituents. Therefore the purpose of this study is to determine the glycemic index of the Fitjoy bar.

ELIGIBILITY:
Inclusion Criteria:

* Participant is between the ages of 18 and 35
* Participant is apparently healthy
* Participant is moderately active and participants in low intensity recreational activity at lease 3 to 4 days a week
* Participant has a BMI < 24.9

Exclusion Criteria:

* Participant has a history of treatment for metabolic disease (i.e., diabetes), hypertension, hypotension, thyroid disease, arrhythmais, cardiovascular disease
* Participant uses current prescription medication (birth control is allowed)
* Participant is pregnant or nursing or plans to become pregnant during the next month
* Participant has an intolerance to caffeine and/or other natural stimulants
* Participant has a history of smoking
* Participant drinks excessively (i.e., 12 drinks per week or more)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
How a commercially available food bar affects blood glucose levels | One day
  Measured in mmol/L
How a commercially available food bar affects blood insulin levels. | One day
  Measured in U/mL

SECONDARY OUTCOMES:
Does a commercially available food bar cause hypoglycemia | One day
  Subjective questionnaire
Does a commercially available food bar cause dizziness | One day
  Subjective questionnaire
Does a commercially available food bar cause headaches | One day
  Subjective questionnaire
Does a commercially available food bar cause fatigue | One day
  Subjective questionnaire
Does a commercially available food bar cause stomach upset | One day
  Subjective questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No